CLINICAL TRIAL: NCT02781441
Title: Evaluation of a Question Prompt List for Patients With Myelodysplastic Syndromes (QPL-MDS)
Acronym: QPL-MDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QPL-MDS-IPC 2014-013
Record Dates: First submitted 2016-05-18; First posted 2016-05-24 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Active Comparator): Patients will receive only the education brochure of GFM
  Interventions: Behavioral: Education brochure of Groupe Français des Myélodysplasies
- General QPL group (Experimental): Patients will receive the brochure and the newly developed QPL (general version)
  Interventions: Behavioral: Question prompt list (QPL); Behavioral: Education brochure of Groupe Français des Myélodysplasies
- Targeted QPL group (Experimental): Patients will receive the brochure and the newly developed QPL (general version)
  Interventions: Behavioral: Question prompt list (QPL); Behavioral: Education brochure of Groupe Français des Myélodysplasies

INTERVENTIONS:
Behavioral: Question prompt list (QPL)
  Arms: General QPL group; Targeted QPL group
Behavioral: Education brochure of Groupe Français des Myélodysplasies

SUMMARY:
MDS are a diverse group of hematopoietic malignancies, which mainly occur in patients over 75 years of age. Incidence rate in 2012 in France was more than 6 cases per 100 000 person-years. MDS are characterized by ineffective haematopoiesis causing cytopenia, and by leukemic transformation. The disease is heterogeneous, its pathophysiology complex and clinical evolution variable.The few data available on MDS patients show how difficult it is to understand MDS, its prognosis and the reasons for prescribing or not some treatments. In the context of a highly complex potentially lethal disease such as MDS, it is of utmost importance to optimize the information conveyed to patients. Particularly, 70.5% of MDS patients surveyed in our developmental study would have preferred more information about prognosis at diagnosis disclosure.

A simple intervention based on the use of a question prompt list (QPL), would greatly improve the information process by helping patients to express their main concerns at their medical consultations. Cultural differences may exist in the appraisal of QPLs and QPLs have not yet been widely used in France.

However, in line with the previous results available in the literature and in a context a priori favourable to the use of such an instrument, the investigators hypothesise that use of a QPL will increase MDS patients' expressions of concerns and questions at their medical consultations. Particularly the investigators assume that the discussion about prognosis will be facilitated, without increasing anxiety because patients remain free to ask or not for such information. The use of QPLs would also be a way to limit social inequalities related to insufficient information and to encourage patient-doctor communication and meeting of patient preferences which could lead to better health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly referred for a MDS in one of the participating centres
* Older than 18
* Able to answer a self-administered questionnaire
* Having signed an informed consent
* affiliated to the French Social Security System

Exclusion Criteria:

* emergency,patients deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Patients having discussed as they wished about the prognosis of their MDS in the next medical consultation | 17 months
  The discussion about prognosis will be collected through the audiotaping of the consultation.

SECONDARY OUTCOMES:
number of questions and concerns expressed in each content category covered by the QPL (including prognosis) | 17 months
  Data collected through the audiotaping of the consultation
Duration of the recorded consultation | 17 months
  Data collected through the audiotaping of the consultation
Quality of life | 17 months
  Questionnaire
Anxiety | 17 months
  Questionnaire
Satisfaction with the provided information | 17 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Rey, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (2):
- France (2):
  - Chu Grenoble, Grenoble
  - Institut Paoli-Calmettes, Marseille

IPD SHARING:
Plan to Share IPD: No